CLINICAL TRIAL: NCT01385449
Title: Continuous Interscalene Block (CISB) Versus Single Injection Interscalene Block in Those Undergoing Shoulder Surgery in the Ambulatory Setting
Brief Title: Prospective Evaluation of Interscalene Nerve Catheters vs. Single Injection Blocks
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: The study was halted prematurely due to low enrollment and anticipation of future barriers to enrollment.
Sponsor: University of Wisconsin, Madison (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: H-2010-0098
Record Dates: First submitted 2011-06-28; First posted 2011-06-30 (Estimated); Last update posted 2019-02-18 (Actual); Status verified 2019-02

CONDITIONS: Pain
Keywords: nerve block; shoulder surgery; physical therapy
MeSH Terms: conditions — Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- interscalene block (Experimental): interscalene block
  Interventions: Procedure: interscalene block
- interscalene catheter (Experimental): interscalene catheter
  Interventions: Procedure: interscalene catheter

INTERVENTIONS:
Procedure: interscalene catheter — interscalene catheter
  Arms: interscalene catheter
Procedure: interscalene block — interscalene block
  Arms: interscalene block

SUMMARY:
The primary hypothesis is that those patients who choose an interscalene catheter will have less pain postoperatively than those with single injection blocks. Secondary hypotheses examine physical therapy outcomes and incidence of parasthesia or pain following surgery for up to 3 months.

ELIGIBILITY:
Inclusion Criteria:

* American Society of Anesthesiologists (ASA) physical status 1-3
* 18-79 years of age, inclusive
* body mass index of < 36 kg/m2.
* The ability to understand local anesthetic related complications and care of a CPNB
* Presence of a caretaker with them during the first 24 hours of local anesthetic infusion, and on a daily basis.
* The ability to communicate with the practitioner managing the catheter.
* Residence within 2 hours of University of Wisconsin Hospital and Clinics

Exclusion Criteria:

* Any contraindication to a continuous interscalene catheter placement
* Clinically significant pulmonary disease
* Clinically significant cardiac disease
* Allergy to ropivacaine
* Peripheral or central nervous system disease
* Current (or planned) anticoagulation therapy or disease
* Local infection over area of catheter placement
* Renal or hepatic failure
* History of opioid dependence
* Significant psychiatric disease
* Pregnancy or lactation (Subjects will be asked if it is possible they could be pregnant. If a subject responds in the affirmative, a pregnancy test will be done.)
* Seizure Disorder

Ages: 18 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 73 (Actual)
Dates: Start 2011-06; Primary Completion 2016-02 (Actual); Study Completion 2016-02 (Actual)

PRIMARY OUTCOMES:
pain on post-operative day 1 | 24 hours
  Pain score on post-operative day 1(POD1) using numeric rating scale (NRS)

SECONDARY OUTCOMES:
Pain post operative day 2 (POD2) | 48 hours
  NRS score on POD2

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - U of Wisconsin, Madison, Wisconsin
  - University of Wisconsin, Madison, Wisconsin